CLINICAL TRIAL: NCT05196945
Title: Vonoprazan Fumarate in Combination With Amoxicillin for the First-line Eradication - a Multicenter, Randomized, Parallel Controlled Study
Brief Title: Vonoprazan Fumarate in Combination With Amoxicillin for the First-line Eradication of Helicobacter Pylori -- a Multicenter, Randomized, Parallel Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Zhejiang University (Other); People's Hospital of Chongqing (Other); Tianjin Medical University General Hospital (Other); Shengjing Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Southern Medical University, China (Other); First People's Hospital of Foshan (Other); Guangzhou Panyu Central Hospital (Other); First Affiliated Hospital of Shantou University Medical College (Other); The Seventh Affiliated Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, pengxiang, Attending physician, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022ZSLYEC-003
Record Dates: First submitted 2022-01-08; First posted 2022-01-19 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori Eradication Rate
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-dual (Experimental): 14 days(vonoprazan fumarate tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 750mg/ time, 4 times/day, oral)
  Interventions: Drug: vonoprazan fumarate + amoxicillin
- EACP - quadruple (Active Comparator): 14days(Esomeprazole 20mg/ time, 2 times/day, oral+Amoxicillin 1g/ time, 2 times/day, oral+Clarithromycin 0.5g/ time, 2 times/day, oral+Bismuth potassium citrate 220mg/ time, twice a day, orally)
  Interventions: Drug: Esomeprazole +Amoxicillin+Clarithromycin+Bismuth potassium citrate

INTERVENTIONS:
Drug: vonoprazan fumarate + amoxicillin — vonoprazan fumarate 20 mg/time, 2 times/day, oral Amoxicillin 750mg/ time, 4 times/day, oral
  Arms: VA-dual
Drug: Esomeprazole +Amoxicillin+Clarithromycin+Bismuth potassium citrate — Esomeprazole 20mg/ time, 2 times/day, oral Amoxicillin 1g/ time, 2 times/day, oral Clarithromycin 0.5g/ time, 2 times/day, oral Bismuth potassium citrate 220mg/ time, twice a day, orally
  Arms: EACP - quadruple

SUMMARY:
Helicobacter pylori infection is closely related to gastritis, peptic ulcer, mucosa-associated lymphoid tissue lymphoma and gastric cancer. Eradication of HP can significantly improve and reduce HP-related diseases. International and domestic guidelines recommend a 10-14 day quadruple regimen containing bismuth as first-line treatment, achieving an eradication rate of more than 80%. However, some disadvantages of these quadruple regimens, such as severe adverse reactions, high medical costs and low compliance, prevent their application in clinical practice. Studies at home and abroad have shown that high-dose proton pump inhibitors combined with amoxicillin can be used as the first-line treatment for HP eradication, with good efficacy and compliance and low rate of adverse reactions. And because it is a single antibiotic therapy, we do not expect this regimen to increase antibiotic resistance rates for HP. The maintenance of gastric PH > 6 is one of the key factors for HP eradication. The acid inhibition effect of proton pump mainly depends on the degree of individual metabolism of proton pump. Vonoprazan fumarate, a new competitive potassium acid blocker, is not affected by gene polymorphism, and has the advantage of stronger and longer inhibition effect on gastric acid compared with proton pump inhibitors. In most parts of China, HP is characterized by high infection rate and antibiotic resistance rate, requiring higher eradication rate and safety regimen. This study compared the efficacy and safety of vonoprazan fumarate combined with amoxicillin and bismuth-containing quadruple regimen in first-line HP eradication, in order to find a more suitable regimen for HP eradication.

ELIGIBILITY:
Inclusion Criteria:

Age 18-70, regardless of gender; HP positive in 13C/14C breath test or pathological test; HP eradication has never been performed in the past; Based on the consensus of helicobacter pylori in 2017, it conforms to the HP eradication guideline; The patient voluntarily signed the informed consent.

Exclusion Criteria:

History of drug allergy in this study; Liver and kidney dysfunction; Cardiopulmonary insufficiency; History of malignant tumor; Taking clopidogrel, warfarin and other drugs simultaneously may affect CYP2C19 metabolism; Pregnant or lactating women; Patients with severe mental illness; Those planning pregnancy; Previous upper gastrointestinal surgery history; Participated in any other clinical investigator in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2022-03-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 6 week
  Rate of h. pylori successfully eradicated；13C-urea breath testthat will be used to assess this outcome measure

SECONDARY OUTCOMES:
Adverse Event | 6 week
  Rate of adverse event, serious adverse event; Questionnaire that will be used to assess this outcome measure.
Medical financial burden | 6 week
  Medical financial burden；Questionnaire that will be used to assess this outcome measure.

IPD SHARING:
Plan to Share IPD: No